CLINICAL TRIAL: NCT04944706
Title: Efficacy and Safety of Qishenyiqi Dripping Pills for Treating Chronic Heart Failure With Preserved Ejection Fraction: a Randomized, Double-blind, Basic-treatment-loading, Placebo-controlled, Multicenter Phase Ⅱ Clinical Trial
Brief Title: Efficacy and Safety of Qishenyiqi Dripping Pills for Treating Chronic Heart Failure With Preserved Ejection Fraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-QSYQDW-HFpEF-Ⅱ
Record Dates: First submitted 2021-06-15; First posted 2021-06-30 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-08

CONDITIONS: Chronic Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — Time

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose group (Experimental): The standard basic treatment is given according to the guidelines related to the underlying disease
  Interventions: Drug: Qishen Yiqi dripping pills 2 bags/time + Qishen Yiqi dripping pills placebo 2 bags/time
- High dose group (Experimental): The standard basic treatment is given according to the guidelines related to the underlying disease
  Interventions: Drug: Qishen Yiqi dripping pills 4 bags/time
- Placebo group (Experimental): The standard basic treatment is given according to the guidelines related to the underlying disease
  Interventions: Drug: Qishen Yiqi dripping pills placebo 4 bags/time

INTERVENTIONS:
Drug: Qishen Yiqi dripping pills 2 bags/time + Qishen Yiqi dripping pills placebo 2 bags/time — Take 3 times a day after meals,24 weeks
  Arms: Low dose group
Drug: Qishen Yiqi dripping pills 4 bags/time — Take 3 times a day after meals,24 weeks
  Arms: High dose group
Drug: Qishen Yiqi dripping pills placebo 4 bags/time — Take 3 times a day after meals,24 weeks
  Arms: Placebo group

SUMMARY:
Main objective: To evaluate the efficacy, safety and clinical dose exploration of Qishen Yiqi dripping pills in the treatment of chronic heart failure with preserved ejection fraction.

DETAILED DESCRIPTION:
Main objective: To evaluate the efficacy, safety and clinical dose exploration of Qishen Yiqi dripping pills in the treatment of chronic heart failure with preserved ejection fraction.

Exploratory research objective: To explore the changes of endogenous substances in vivo before and after drug administration, to interpret the mechanism of drug action through metabolomics and systems biology methods, and to find potential clinical biomarkers for exploratory subgroup analysis of clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥ 18 years
* Diagnosed as chronic heart failure with preserved ejection fraction according to the Guidelines for Diagnosis and Treatment of Heart Failure in China 2018

  1. Have symptoms and/or signs of chronic heart failure at least 30 days before the trial
  2. LVEF≥50% according to echocardiography during screening stage
  3. BNP > 35 ng/L and/or NT-proBNP > 125 ng/L
  4. Cardiac structural changes or diastolic dysfunction according to echocardiography during screening stage, in line with at least one of the following:

     1. : LAVI>34ml/m2
     2. : E/e'≥13
     3. : average e'(interventricular septum and free wall)<9cm/s
* NYHAⅡ-Ⅲ
* Patients with hypertension received a stable dose of antihypertensive therapy for at least 4 weeks and kept their blood pressure at an ideal level for at least 4 weeks
* Ability to understand the requirements of the study and willingness to provide written informed consent
* Have no pregnancy program and take effective contraceptive measures voluntarily
* Abide by the experimental protocol and cooperate with the data collection according to the researcher's judgment

Exclusion Criteria:

* People with any of the following cardiovascular diseases:

  1. Patients with acute decompensated heart failure who need to use quick-acting diuretics, vasodilators, or positive inotropic drugs for treatment, or in the adjustment period of acute decompensated heart failure treatment, and the adjustment time is less than 1 month
  2. Clinical evidence of acute coronary syndrome (including myocardial infarction, unstable angina pectoris) within 6 months before screening stage
  3. Received prior revascularization (such as PCI, CABG), or implantable cardioverter defibrillator (ICD), or other cardiac/cardiovascular procedures within 3 months before screening stage
  4. Received cardiac resynchronization therapy (CRT) within 6 months before screening stage
  5. Implantable devices (e.g. ICD, CRT), revascularization (e.g. PCI, CABG), or other cardiac/cardiovascular procedures are expected to be performed during the trial period
  6. Patients with acute myocarditis, invasive cardiomyopathy, constrictive pericarditis, cardiac tamponade, hypertrophic obstructive cardiomyopathy, cardiac shock, hemodynamic abnormalities of heart valve disease significantly narrow and/or regurgitation (moderate or above, etc.), Ⅱ degrees above Ⅱ type atrioventricular block placement pacemaker therapy, average QTc > 450 ms or heart rate < 50 times/min
  7. Patients with pulmonary artery embolism caused by pulmonary hypertension, chronic obstructive pulmonary disease and other serious pulmonary diseases
  8. Hypertension that is difficult to control with medication (systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg)
  9. Symptomatic hypotension and/or systolic blood pressure <100 mmHg
* Severe renal insufficiency: eGFR < 30 ml/min/1.73m2
* ALT and AST > 3 times upper the limit of normal values in local laboratories, and/or total bilirubin > 2 times upper the limit of normal values in local laboratories
* Serum potassium ≥5.5 mmol/L
* HbA1c≥9.0%, or fasting blood glucose >13.9 mmol/L
* Diabetic patients who are using sodium-glucose cotransporter 2 inhibitors and cannot stop using them during the trial, such as dagliredin, entagliredin, and cagliredin
* The ECG examination indicated the onset of atrial fibrillation during the screening period or previous history of atrial fibrillation within 6 months before screening stage
* Hemoglobin < 9.0 g/dL
* Patients have stroke 3 months before the screening period
* Concomitant mental illness and poor condition control, which affects the signing of informed consent or presentation of adverse events
* Patients with active malignancies (including those currently under oncology treatment)
* Unable to conduct the 6-minute walking distance test due to physical impairment or other non-cardiac reasons
* Women who are pregnant or lactating
* Allergic constitution, or allergic to the test drug or its ingredients
* Participate in clinical trials of other drugs within 3 months before screening
* The researchers did not consider it appropriate to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
6-Minutes-Walking-Test (6MWT) | Baseline to weeks 12 and 24
  Change from baseline to weeks 12 and 24 in exercise capacity as measured by the 6-Minutes-Walking-Test (6MWT) distance.

SECONDARY OUTCOMES:
NT-proBNP | Baseline to weeks 2,4,8,12,16,20 and 24
  Change from baseline to weeks 2,4,8,12,16,20 and 24 in NT-proBNP.
LAVI, E/ E ', E 'mean value, LVEF and tricuspid regurgitation velocity | Baseline to weeks 4,12 and 24
  Change from baseline to weeks 4,12 and 24 in left atrial volume index, mitral inflow velocity early diastolic blood flow velocity peak to mitral annular relaxation velocity ratio, mitral annular relaxation velocity mean value, left ventricular ejection fraction and tricuspid regurgitation velocity measured by echocardiography.
Hospitalizations for heart failure (first or repeated) and deaths from cardiovascular disease | Week 24
  Compound and separate rates of hospitalization for heart failure (first or repeated) and death from cardiovascular disease at week 24.
NYHA classification | Baseline to weeks 2,4,8,12,16,20 and 24
  Percentage of subjects whose NYHA classification improved/worsened/remained unchanged from baseline to weeks 2,4,8,12,16,20 and 24.
Minnesota Living With Heart Failure Questionnaire(MLHFQ) Score | Baseline to weeks 12 and 24
  Change from baseline to weeks 12 and 24 in Minnesota Living With Heart Failure Questionnaire(MLHFQ) Score.

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Bejing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The Third Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan
  - The third Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - China Japan Union Hospital of Jilin University, Changchun, Jilin
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Nei Monggol Autonomous Region
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Second Affiliated Hospital Of Xi'an Jiaotong University, Xi’an, Shanxi
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality